CLINICAL TRIAL: NCT07209293
Title: The Effect of Orogastric Suctioning on Quality of Transesophageal Echo Images in Cardiac Surgery
Brief Title: Oral Gastric Suctioning Effect on Transesophageal Echo
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00137024
Record Dates: First submitted 2025-09-30; First posted 2025-10-06 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-09

CONDITIONS: TEE Image Quality
Keywords: gastric suction; transesophageal echocardiography; cardiac surgery
MeSH Terms: interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cardiac Surgery with Transesophageal Echocardiography: Participants scheduled for cardiac surgery with transesophageal echocardiography performed as part of their standard of care treatment during their surgery.
  Interventions: Diagnostic Test: Transesophageal Echocardiography

INTERVENTIONS:
Diagnostic Test: Transesophageal Echocardiography — Transesophageal echocardiography images will be taken prior to and post oral gastric suction.

SUMMARY:
During heart surgery images of the heart are taken with transesophageal echocardiography. The images track how the heart is doing during surgery. It is normal practice to place an oral gastric tube in the stomach during heart surgery. The oral gastric tube is used to suction out stomach contents to avoid potential aspiration and avoid stomach acid build up. The purpose of this research study is to see if the images of the heart have better quality after your stomach has been emptied. This project hopes to help determine the best method to obtain the better quality images of the heart during cardiac surgery.

DETAILED DESCRIPTION:
After induction, the transesophageal echocardiography (TEE) probe will be placed in the usual fashion for the cardiac surgery case. Five specific images that are part of a standard TEE exam will be obtained by TEE. An oral gastric (OG) tube will then be placed to suction stomach contents. The OG tube will then be removed and the same five images previously taken will be repeated. The five images reviewed from the TEE include mid esophageal four chamber, mid esophageal two chamber, transgastric basal, transgastric mid-papillary and deep transgastric. Two blinded and independent cardiologists who are echocardiography experts will review the before and after images and grade them for quality of the images. They will grade the images on a scale of 1-4 with 1 being excellent quality and 4 being very poor quality.

ELIGIBILITY:
Inclusion Criteria:

- Transesophageal echocardiography assisted cardiac surgery

Exclusion Criteria:

* hiatal hernia
* documented or suspected esophageal stricture
* contraindications to a TEE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for cardiac surgery at Atrium Health Wake Forest Baptist
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Mid Esophageal Four Chamber Images - Pre Oral Gastric Suction | 60 minutes
  Using transesophageal echocardiography mid esophageal four chamber images will be taken prior to oral gastric suctioning. Quality of images will be graded on a scale of 1-4 (1=excellent quality, 4=very poor quality).
Quality of Mid Esophageal Four Chamber Images - Post Oral Gastric Suction | 60 minutes
  Using transesophageal echocardiography mid esophageal four chamber images will be taken post oral gastric suctioning. Quality of images will be graded on a scale of 1-4 (1=excellent quality, 4=very poor quality).
Quality of Transgastric Basal Images - Pre Oral Gastric Suction | 60 minutes
  Using transesophageal echocardiography transgastric basal images will be taken prior to oral gastric suctioning. Quality of images will be graded on a scale of 1-4 (1=excellent quality, 4=very poor quality).
Quality of Transgastric Basal Images - Post Gastric Suction | 60 minutes
  Using transesophageal echocardiography transgastric basal images will be taken post oral gastric suctioning. Quality of images will be graded on a scale of 1-4 (1=excellent quality, 4=very poor quality).
Quality of Transgastric Mid Papillary Images - Pre Oral Gastric Suction | 60 minutes
  Using transesophageal echocardiography transgastric mid images will be taken prior to oral gastric suctioning. Quality of images will be graded on a scale of 1-4 (1=excellent quality, 4=very poor quality).
Quality of Transgastric Mid Papillary Images - Post Oral Gastric Suction | 60 minutes
  Using transesophageal echocardiography transgastric mid images will be taken post oral gastric suctioning. Quality of images will be graded on a scale of 1-4 (1=excellent quality, 4=very poor quality).
Quality of Mid Esophageal Two-Chamber Images - Pre Oral Gastric Suction | 60 minutes
  Using transesophageal echocardiography mid esophageal two-chamber images will be taken prior to oral gastric suctioning. Quality of images will be graded on a scale of 1-4 (1=excellent quality, 4=very poor quality).
Quality of Mid Esophageal Two-Chamber Images - Post Oral Gastric Suction | 60 minutes
  Using transesophageal echocardiography mid esophageal two-chamber images will be taken post oral gastric suctioning. Quality of images will be graded on a scale of 1-4 (1=excellent quality, 4=very poor quality).
Quality of Deep Transgastric Images - Pre Oral Gastric Suction | 60 minutes
  Using transesophageal echocardiography deep transgastric images will be taken prior to oral gastric suctioning. Quality of images will be graded on a scale of 1-4 (1=excellent quality, 4=very poor quality).
Quality of Deep Transgastric Images - Post Oral Gastric Suction | 60 minutes
  Using transesophageal echocardiography deep transgastric images will be taken post oral gastric suctioning. Quality of images will be graded on a scale of 1-4 (1=excellent quality, 4=very poor quality).

CONTACTS AND LOCATIONS:
Overall Officials: Scott Coleman, DO, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health-Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No